CLINICAL TRIAL: NCT00723996
Title: Preventive Health Behavior in Women
Status: Completed | Type: Observational
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Ruth Carlos M.D., Principal Investigator, University of Michigan
Other Study IDs: HUM00048680
Record Dates: First submitted 2008-07-24; First posted 2008-07-29 (Estimated); Last update posted 2016-12-16 (Estimated); Status verified 2016-12

CONDITIONS: Colon Cancer
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Group 1: Women receiving a CRC-related questionnaire and a CRC educational video.
  Interventions: Behavioral: Behavioral Study in Women
- Group 2: Women who receive only a CRC-related questionnaire.
- Group 3: Women who receive neither questionnaire nor educational video.
  Interventions: Behavioral: Behavioral Study in Women

INTERVENTIONS:
Behavioral: Behavioral Study in Women — A Randomized study to assess the knowledge of womens health related issues
  Groups: Group 1; Group 3

SUMMARY:
The overall goal of the proposed research is to explore behavioral correlations between colorectal cancer screening and screening mammography.

DETAILED DESCRIPTION:
The overall goal of the proposed research is to explore behavioral correlations between colorectal cancer screening and screening mammography and to develop an innovative approach for reducing barriers colorectal cancer screening in women, using screening mammography, an existing non-colon cancer related screening test that has widespread public acceptance, as a "teachable moment." Although screening for colorectal cancer (CRC) has been shown to decrease the incidence of CRC and CRC associated mortality, adherence to screening guidelines from the American Cancer Society and the American Gastroenterological Association remains poor.1-5 Barriers to adherence are not fully defined, but may include poor understanding of the relative benefits and risks of CRC screening, absence of physician recommendation, lack of insurance coverage for screening procedures, and poor patient acceptance of screening procedures. A potential challenge in increasing patient knowledge may be the milieu in which the educational intervention is administered. This study will be the first prospective study to evaluate the effectiveness of an educational intervention designed to increase CRC screening administered at a cancer screening visit unrelated to CRC.

ELIGIBILITY:
Inclusion Criteria:

1. Women between the ages of 50 and 75 years old.
2. Scheduled for a screening mammogram.

Exclusion Criteria:

1. CRC screening current (FOBT within preceding 12 months, FS within 5 years, or colonoscopy within 10 years).
2. Family history of CRC in a first-degree relative.
3. Personal history of colonic adenomatous polyps, CRC or inflammatory bowel disease

Ages: 50 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Women who are scheduled for a screening mammogram at a University Medical Center who are between 50 and 75 years old will recruited.
Sampling Method: Non-Probability Sample
Enrollment: 254 (Actual)
Dates: Start 2003-09; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
The primary outcome will be determined through review of medical records or a telephone follow-up 6 months after enrollment | At 6 month intervals

CONTACTS AND LOCATIONS:
Overall Officials: Ruth Carlos, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan Health System, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No